CLINICAL TRIAL: NCT01824888
Title: The Effectiveness and Efficacy of Using JUC Antimicrobial Spray for Controlling the Infection Transmission
Brief Title: Efficacy of JUC as Hand Rub Evaluated by Using European Standard 1500
Acronym: JUC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, John Yuen, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: JUC-001-EN1500; 8-ZDA4 (Other Grant/Funding Number: PolyU-Grant-8-ZDA4)
Record Dates: First submitted 2013-03-22; First posted 2013-04-05 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Infectious Disease Transmission
Keywords: JUC; hand rub; European standard
MeSH Terms: interventions — 2-Propanol; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Following standard one-minute handwashing, both hands were immersed up to the mid-metacarpals for 5 seconds into a contamination fluid containing E. coli. Handrubs were performed by using 60% propan-2-ol into the cupped hands and rub vigorously for 30 seconds, the procedure was completed by a 5 seconds rinse of the fingers under running tap water and excess water was shaken off.
  Interventions: Drug: propan-2-ol
- JUC solution (Experimental): Following standard one-minute handwashing, both hands were immersed up to the mid-metacarpals for 5 seconds into a contamination fluid containing E. coli. Handrubs were performed by pouring 1.5 ml of JUC into the cupped hands and rub vigorously for 30 seconds, the procedure was completed by a 5 seconds rinse of the fingers under running tap water and excess water was shaken off.
  Interventions: Drug: JUC solution

INTERVENTIONS:
Drug: JUC solution — 1.5 ml JUC solution rubbing on hands for 30 seconds, repeated twice
  Other Names: JUC physical antimicrobial dressing
  Arms: JUC solution
Drug: propan-2-ol — 1.5 ml propan-2-ol rubbing on hands for 30 seconds, repeated twice
  Other Names: alcohol reference
  Arms: Control

SUMMARY:
JUC is a commercially available wound care spray. It is evaluated for the efficacy when using as a hygienic hand rub following the protocol described in the European standard EN 1500:1997 "Chemical disinfectants and antiseptics - Hygienic handrub - Test method and requirement (phase 2/step 2)". A crossover study to compare the JUC solution with 60% (v/v) propan-2-ol by using Escherichia coli K12 NCTC strain 10538 as test organism.

DETAILED DESCRIPTION:
Before the intervention, the bactericidal activity of JUC was validated in accordance with the prEN 12054. A total of 15 volunteers were recruited, hands were washed immediately prior to the intervention. Then, both hands of each volunteer were immersed into a contamination fluid of E. coli. Then, hand rub was performed with JUC or alcohol. Culture samples were collected before and after the hand rub by rubbing the fingertips and thumb tips of each hand ont he base of a Petri dish containing appropriate medium. The culture inoculation, incubation, appropriate dilutions, and colony count were performed.

ELIGIBILITY:
Inclusion Criteria:

* healthy and absence of significant illness

Exclusion Criteria:

* Visible wounds on hands

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change of Colony forming units on hands from pre-value (baseline) to post-value | Pre-value (baseline) as 0 minutes: at the time after handwashing and before application of JUC or alcohol; Post-value at 5 minutes after the baseline: as after hand contamination, application of JUC or alcohol and drying of hands
  Pre-value and post-value were collected by rubbing the fingertips and thumb tips of each hand for 1 minute on the base of a Petri dish containing medium. Then the samples with appropriate dilutions were plated onto agar plates for incubation, and colony forming units of the plates were counted.

SECONDARY OUTCOMES:
Change of colony forming units on hands from baseline to 8 hours after hand rubbing with JUC | Pre-value (baseline) at 0 hour: at the first time after applicaiton of JUC and challenged by the bacteria; Post-values measured at each hour (1,2,3,4,5,6,7 and 8 hours) after the initial application of JUC and bacterial challenge at every hour
  JUC was applied after handwashing, an invisible protective frame will be formed on treated hands. Samples were collected for culture each hour after the challenge of the E. coli contamination fluid.Pre-value and post-value were collected by rubbing the fingertips and thumb tips of each hand for 1 minute on the base of a Petri dish containing medium. Then the samples with appropriate dilutions were plated onto agar plates for incubation, and colony forming units of the plates were counted.

OTHER OUTCOMES:
Bactericidal efficacy of JUC and neutralizer | 1 day
  Mixing the JUC with or without neutralizer with a fixed amount of E. coli to assess the bactericidal effects.

CONTACTS AND LOCATIONS:
Overall Officials: John Yuen, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- PolyU Biomedical Science Laboratory, Kowloon, Hong Kong